CLINICAL TRIAL: NCT03656809
Title: Feasibility of Multi-gene Panel Testing at the Time of Diagnosis for Patients With Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01459
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — multi-gene panel testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the feasibility of routine referral to genetic counseling for all patients with a new diagnosis of epithelial ovarian, primary peritoneal or fallopian tube cancer.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have a new diagnosis of epithelial ovarian, primary peritoneal, fallopian tube or extra- uterine mullerian cancer.
* All subjects must have either undergone primary surgery or be planning neoadjuvant chemotherapy for the treatment of ovarian, primary peritoneal or fallopian tube cancer.
* All subjects must be able to comprehend and communicate in English.
* All subjects must agree to participate.
* A previous diagnosis of cancer is not an exclusion criterion.
* Previous genetic screening is not an exclusion criterion.

Exclusion Criteria:

* Patients who do not meet the above inclusion criteria.
* Patients with a diagnosis of a low malignant potential mullerian tumor.
* Patients who are not proficient in English language because the survey aspect of this study is comprised of 4 validated surveys that are only available in English language.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females with ovarian cancer
Study Population: new diagnosis of epithelial ovarian, primary peritoneal, fallopian tube or extra- uterine mullerian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of timely routine referral to genetic counseling for all patients with a new diagnosis of epithelial ovarian, primary peritoneal or Fallopian tube cancer. | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Levine, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States